CLINICAL TRIAL: NCT02739035
Title: Manipulation Under Anesthesia (MUA) to Treat Postoperative Stiffness After Total Knee Arthroplasty: A Multicenter Randomized Clinical Trial
Brief Title: MUA to Treat Postoperative Stiffness After Total Knee Arthroplasty
Acronym: MUA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Knee Society (Other)
Responsible Party: Principal Investigator, Matthew P. Abdel, M.D., Consultant - Knee Surgery, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-009075
Record Dates: First submitted 2016-03-31; First posted 2016-04-14 (Estimated); Results first posted 2023-11-21 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Stiffness Following Total Knee Arthroplasty
MeSH Terms: interventions — Dexamethasone; Calcium Dobesilate; Celecoxib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MUA alone (No Intervention): Subjects will be given manipulation under anesthesia, will fill out questionnaires about their knee and quality of life and will be followed throughout their routine follow up to assess their continued process. Subjects will fill out questionnaires at the time of their consent and their 6-week and 1-year follow up visits. The questionnaires will take about 15-20 minutes to complete.
- MUA with dexamethasone and celecoxib (Experimental): For subjects assigned to the MUA with anti-inflammatory medication group, an intravenous (into the vein) dose of dexamethasone will be given at the time of MUA. Subjects in this group will also receive celecoxib. They will be asked to take the medicine one time daily either at morning or night time with food and water for 2 weeks following MUA. Subjects will also be followed throughout their routine follow up to assess their continued process, and they will fill out questionnaires at the time of their consent and their 6-week and 1-year follow up visits. The questionnaires will take about 15-20 minutes to complete.
  Interventions: Drug: Dexamethasone; Drug: Celecoxib

INTERVENTIONS:
Drug: Dexamethasone — 8 mg of IV dexamethasone immediately before MUA.
  Other Names: Decadron
  Arms: MUA with dexamethasone and celecoxib
Drug: Celecoxib — 2 weeks per mouth of celecoxib (200 mg daily)
  Other Names: Celebrex
  Arms: MUA with dexamethasone and celecoxib

SUMMARY:
Compare the outcome following manipulation under anesthesia for stiffness in a randomized controlled fashion with one group receiving IV dexamethasone and oral celecoxib at the time of manipulation to a control group receiving manipulation alone.

Outcomes will include pain, range of motion, as well as subjective outcome scores.

DETAILED DESCRIPTION:
Stiffness is a potential complication following Total Knee Arthroplasty (TKA). While a variety of factors have been cited as possible causes, such as component malrotation or improper soft-tissue balancing, however, an etiology is not always appreciated. Histologic and arthroscopic evidence of fibrosis suggests that an inflammatory process may contribute to loss of knee range of motion following surgery. Manipulation under anesthesia remains standard of care for stiffness following TKA. Manipulation shows improved range of motion for stiffness after total knee arthroplasty, however, patients do not always achieve full range of motion. Furthermore, repeat manipulation and manipulation greater than 8 weeks post-surgically have shown limited improvements. Given a possible role of the host inflammatory response and the importance of early gains in knee range of motion following total knee arthroplasty, limiting the inflammatory response at the time of manipulation may improve outcomes. Investigators would like to assess the role of anti-inflammatory medications to optimize range of motion and outcome for manipulation under anesthesia for stiffness following TKA.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who have received a primary unilateral TKA for a diagnosis of osteoarthritis.
2. MUA's scheduled between 6-10 weeks postoperatively

Exclusion Criteria:

1. Intolerance to NSAIDs
2. Renal dysfunction
3. Age < 18 or > 90 years
4. Primary diagnosis of rheumatoid arthritis
5. Patients with a Glomerular Filtration Rate (GFR) <60 as the cut off for Chronic Kidney Disease (CKD) (stage 3 CKD)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2022-12 (Actual); Study Completion 2022-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Abdel Matthew, M.D., Principal Investigator — Mayo Clinic
Locations (16):
- United States (16):
  - HipKnee Arkansas Foundation, Little Rock, Arkansas
  - Colorado Joint Replacement, Denver, Colorado
  - Rush University Medical Center, Chicago, Illinois
  - Mayo Clinic, Rochester, Minnesota
  - Univ. of Nebraska Medical Center, Omaha, Nebraska
  - Hospital for Joint Diseases, New York, New York
  - Hospital for Special Surgery, New York, New York
  - New York - Presbyterian at Columbia University, New York, New York
  - OrthoCarolina, Charlotte, North Carolina
  - Duke University Medical Ceter, Dept. of Orthopaedics, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Joint Implant Surgeons, New Albany, Ohio
  - Rothman Institute, Lansdale, Pennsylvania
  - Aria 3B Orthopaedic Specialists, Philadelphia, Pennsylvania
  - Houston Methodist, Houston, Texas
  - University of Utah Orthopaedic Center, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 16 orthopedic surgery centers across the United States. Enrollment took place between 2016 and 2021. The first patient was enrolled in October of 2016 and the final patient was enrolled in November of 2021.
Pre-assignment Details: 441 patients were screened for eligibility, 130 of which met inclusion criteria, were enrolled in the trial and had treatment randomization.
Period: 6 Weeks Post-MUA
Arm/Group | MUA Alone | MUA With Dexamethasone and Celecoxib
Started | 59 | 71
Completed | 56 | 61
Not Completed | 3 | 10
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Lost to Follow-up | 1 | 3
Not completed — Protocol Violation | 1 | 4
Period: 1 Year Post-MUA
Arm/Group | MUA Alone | MUA With Dexamethasone and Celecoxib
Started | 56 | 61
Completed | 46 | 50
Not Completed | 10 | 11
Not completed — Lost to Follow-up | 10 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MUA Alone | MUA With Dexamethasone and Celecoxib | Total
Number analyzed (Participants) | 59 | 71 | 130
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.6 (10.9) | 61.8 (8.4) | 61.7 (9.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 48 | 82
  Male | 25 | 23 | 48
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Weight (kg) [Mean (Standard Deviation); unit: kilograms] | 90.0 (18.0) | 88.6 (19.6) | 89.3 (18.8)
Height (cm) [Mean (Standard Deviation); unit: centimeters] | 169.2 (10.4) | 166.6 (11.0) | 167.9 (10.7)
BMI (kg/m^2) [Mean (Standard Deviation); unit: Kilograms per meter-squared] | 31.4 (5.6) | 32.2 (6.0) | 31.8 (5.8)
ASA Status (n, %) [Count of Participants; unit: Participants] — The American Society of Anesthesiologists Physical Status Classification System (ASA Status) contains 6 total categories for assessing the physical health of patients.
  Class I: Healthy person Class II: Mild systemic disease (i.e. controlled diabetes or minor infection) Class III: Severe systemic disease ( Class IV: Life threatening systemic disease Class V: Moribund and is not expected to survive without operation Class VI: Declared brain dead, but donating organs
  For the purposes of this study, only patients from classes I-IV were enrolled.
  Participants
    I | 4 | 5 | 9
    II | 39 | 46 | 85
    III | 13 | 17 | 30
    IV | 1 | 0 | 1
    Unknown | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Knee Range of Motion After Manipulation Under Anesthesia
Description: Knee range of motion after manipulation will be measured in degrees as the total arc of motion from maximum passive flexion to maximum passive extension.
Time Frame: 6 weeks after manipulation
Population: Patients who were able to complete follow-up and have range of motion measured.
Measure: Mean (Full Range); unit: Degrees
Arm/Group | MUA Alone | MUA With Dexamethasone and Celecoxib
Number analyzed (Participants) | 53 | 58
Degrees | 98.7 [60 to 125] | 101.2 [75 to 124]
Statistical Analysis 1: Comparison: MUA Alone vs MUA With Dexamethasone and Celecoxib; Outcomes were compared between the two study groups using two-sample t-tests. T-tests were two-sided and the standard alpha value of 0.05 was the threshold for statistical significance. The null hypothesis was that there were no significant differences between control group of MUA alone and the treatment group of MUA with dexamethasone and celecoxib; Test type: Superiority — A difference of 10 degrees in total mean range of motion between the control and the treatment group was considered a clinically significant improvement; p = 0.23, t-test, 2 sided — Using a standard alpha value of 0.05, p values below 0.05 were considered statistically significant

2. Primary Outcome: Knee Range of Motion After Manipulation Under Anesthesia
Description: as for outcome 1
Time Frame: 1 year from the date of the manipulation
Population: Patients who were able to complete a follow-up at the 1-year mark and have knee range of motion measured.
Measure: Mean (Full Range); unit: Degrees
Arm/Group | MUA Alone | MUA With Dexamethasone and Celecoxib
Number analyzed (Participants) | 38 | 45
Degrees | 107.7 [54 to 135] | 107.6 [70 to 130]
Statistical Analysis 1: Comparison: MUA Alone vs MUA With Dexamethasone and Celecoxib; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — A difference of 10 degrees in total mean range of motion (ROM) between the control and the treatment group was considered a clinically significant improvement. To detect this difference, a previous study's mean and standard deviation were referenced in order to predict the variation of results. 54 patients per arm were required to have 90% power with a two-sided t-test and a type I error rate of 5%. 130 patients were targeted for recruitment to account for up to a 20% dropout rate; p = 0.81, t-test, 2 sided — Using a standard alpha value of 0.05, p values below 0.05 were considered statistically significant

3. Secondary Outcome: Knee Society Functional Score
Description: The Knee Society Functional score was developed by the Knee Society as a method of evaluating how well a patient can use their joint. Knee function was evaluated in two categories: walking, and stair usage. Points range from 0-100. 0 = extreme problems, 100 = no problems.
  In each category, points range from 0-50, where 0 = extreme problems to 50 = no problems. Total scores are 0-100 with lower scores indicating extreme knee function problems and higher scores indicating no knee function problems.
Time Frame: 6 weeks after the MUA, and 1 year after the MUA
Population: Patients who were able to complete and return KSS Functional surveys.
Measure: Mean (Standard Deviation); unit: score on a 0-100 scale
Arm/Group | MUA Alone | MUA With Dexamethasone and Celecoxib
Number analyzed (Participants) | 53 | 59
score on a 0-100 scale
  6 weeks after MUA | 64.7 (22.5) | 64.2 (19.2)
  1 year after MUA: number analyzed (Participants) | 40 | 44
  1 year after MUA | 77.3 (24.9) | 74.2 (20.8)

4. Secondary Outcome: Knee Society Knee Score
Description: The Knee Society Knee Score is method of joint evaluation developed by the Knee Society to measure the condition of a patient's knee. Knee condition was evaluated in three categories: pain, range of motion, and stability. Points range from 0-100. 0 = extreme problems, 100 = no problems.
  Up to 50 points for pain, 25 points for range of motion, and 25 points for stability. Deductions occur for Extension lag, flexion contracture, malalignment, and pain at rest.
Time Frame: 6 weeks after the MUA, and 1 year after the MUA
Population: Patients who were able to complete and return the KSS survey.
Measure: Mean (Standard Deviation); unit: Score on a 0-100 scale
Arm/Group | MUA Alone | MUA With Dexamethasone and Celecoxib
Number analyzed (Participants) | 52 | 58
Score on a 0-100 scale
  6 weeks after MUA | 65.1 (17.6) | 66.8 (16.9)
  1 year after MUA: number analyzed (Participants) | 35 | 39
  1 year after MUA | 74.2 (16.1) | 68.6 (24.9)

5. Secondary Outcome: Short Form Survey 12-item Version 2 (SF-12v2): Physical Health
Description: The SF-12v2 questionnaire uses questions selected from the longer SF-36 Health Survey to measure patient wellness and quality of life. Responses were scored using the SF12v2 New England Medical Center (NEMC) scoring algorithm which converts the raw score from the questionnaire into a t-score. The algorithm is calibrated so that an average healthy person would have a t-score of 50 points with a standard deviation of 10. Higher scores indicate better physical health.
Time Frame: 6 weeks after the MUA, and 1 year after the MUA
Population: Patients who were able to complete and return the Physical Health portion of the SF-12 survey.
Measure: Mean (Standard Deviation); unit: t-score
Arm/Group | MUA Alone | MUA With Dexamethasone and Celecoxib
Number analyzed (Participants) | 54 | 60
t-score
  6 weeks after MUA | 38.7 (9.4) | 37.0 (9.7)
  1 year after MUA: number analyzed (Participants) | 40 | 44
  1 year after MUA | 44.8 (10.8) | 43.3 (10.3)

6. Secondary Outcome: Short Form Survey 12-item Version 2 (SF-12v2): Mental Health
Description: The SF-12v2 questionnaire uses questions selected from the longer SF-36 Health Survey to measure patient wellness and quality of life. Responses were scored using the SF12v2 New England Medical Center (NEMC) scoring algorithm which converts the raw score from the questionnaire into a t-score. The algorithm is calibrated so that an average healthy person would have a t-score of 50 points with a standard deviation of 10. Higher scores indicate better mental health.
Time Frame: 6 weeks after MUA, 1 Year after MUA
Population: Patients who completed and returned the SF-12 survey.
Measure: Mean (Standard Deviation); unit: t-score
Arm/Group | MUA Alone | MUA With Dexamethasone and Celecoxib
Number analyzed (Participants) | 54 | 60
t-score
  6 weeks after MUA | 51.7 (9.9) | 53.7 (9.8)
  1 year after MUA: number analyzed (Participants) | 40 | 44
  1 year after MUA | 54.4 (8.8) | 54.3 (8.9)

7. Secondary Outcome: Knee Injury and Osteoarthritis Outcome Score (KOOS): Symptom Score
Description: The KOOS is a commonly used questionnaire which focuses on how patients are affected by osteoarthritis symptoms in five areas: knee pain, stiffness, daily activity, sport and recreation, and quality of life. Results are scored 0-100. 0 = extreme problems, 100 = no problems.
Time Frame: 6 weeks after the MUA, and 1 year after the MUA
Population: Patients who completed the KOOS questionnaire and returned it.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | MUA Alone | MUA With Dexamethasone and Celecoxib
Number analyzed (Participants) | 16 | 17
Score on a scale
  6 weeks after MUA | 64.2 (22.4) | 58.0 (19.9)
  1 year after MUA: number analyzed (Participants) | 10 | 15
  1 year after MUA | 82.5 (11.0) | 75.7 (16.0)

8. Secondary Outcome: Knee Injury and Osteoarthritis Outcome Score (KOOS): Pain Score
Description: as for outcome 7
Time Frame: 6 weeks after the MUA, and 1 year after the MUA
Population: Patients who completed the KOOS survey and returned it.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | MUA Alone | MUA With Dexamethasone and Celecoxib
Number analyzed (Participants) | 17 | 17
Score on a scale
  6 weeks after MUA | 68.9 (20.3) | 62.7 (18.1)
  1 year after MUA: number analyzed (Participants) | 11 | 15
  1 year after MUA | 84.1 (10.7) | 79.8 (17.0)

9. Secondary Outcome: Knee Injury and Osteoarthritis Outcome Score (KOOS): Activities of Daily Living (ADL) Score
Description: as for outcome 7
Time Frame: 6 weeks after MUA, 1 year after MUA
Population: Patients who completed and returned the KOOS survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MUA Alone | MUA With Dexamethasone and Celecoxib
Number analyzed (Participants) | 16 | 17
score on a scale
  6 weeks after MUA | 74.1 (13.7) | 70.3 (16.4)
  1 year after MUA: number analyzed (Participants) | 11 | 15
  1 year after MUA | 81.0 (18.1) | 76.6 (20.6)

10. Secondary Outcome: Knee Injury and Osteoarthritis Outcome Score (KOOS): Sport and Recreation Score
Description: as for outcome 7
Time Frame: 6 weeks after MUA, 1 year after MUA
Population: Patients who completed the KOOS survey and returned it.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MUA Alone | MUA With Dexamethasone and Celecoxib
Number analyzed (Participants) | 8 | 10
score on a scale
  6 weeks after MUA | 48.5 (21.0) | 52.8 (17.7)
  1 year after MUA: number analyzed (Participants) | 7 | 10
  1 year after MUA | 61.0 (25.3) | 62.2 (19.8)

11. Secondary Outcome: Knee Injury and Osteoarthritis Outcomes Score (KOOS): Quality of Life
Description: as for outcome 7
Time Frame: 6 weeks after MUA, 1 year after MUA
Population: Patients who completed the KOOS survey and returned it.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MUA Alone | MUA With Dexamethasone and Celecoxib
Number analyzed (Participants) | 16 | 17
score on a scale
  6 weeks after MUA | 49.2 (22.2) | 50.0 (22.8)
  1 year after MUA: number analyzed (Participants) | 11 | 15
  1 year after MUA | 83.0 (12.8) | 67.1 (27.2)

12. Secondary Outcome: Knee Injury and Osteoarthritis Outcome Score (KOOS) for Joint Replacement (JR)
Description: KOOS JR is a questionnaire designed to measure outcomes for patients with knee replacements. Questions focus on knee stiffness, pain, and function for daily activities. Results are scored 0-100. 0 = extreme problems, 100 = no problems.
Time Frame: 6 weeks after the MUA, and 1 year after the MUA
Population: Patients who completed the KOOS JR survey and returned it.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MUA Alone | MUA With Dexamethasone and Celecoxib
Number analyzed (Participants) | 44 | 53
score on a scale
  6 weeks after MUA | 64.9 (17.7) | 62.7 (13.1)
  1 year after MUA: number analyzed (Participants) | 41 | 43
  1 year after MUA | 72.5 (17.0) | 69.0 (18.9)

13. Secondary Outcome: PROMIS-29 Outcome Form: Physical Function
Description: The PROMIS-29 outcome form measures physical and mental health outcomes for patients. Patients responded to 29 questions in seven categories: physical function, pain interference, depressive symptoms, anxiety, ability to participate in social activities, and sleep disturbance. Scores were scaled so that an average healthy person would score 50 points. A higher score represents more of what is being measured. For physical function, higher scores indicate better function.
  Patient questionnaire responses are scored using the PROMIS-29 scoring algorithm. Scores are scaled to a mean of 50 for a healthy reference population with a standard deviation of 10.
Time Frame: 6 weeks after the MUA, and 1 year after the MUA
Population: Patients who completed the PROMIS-29 survey and returned it.
Measure: Mean (Standard Deviation); unit: t-score
Arm/Group | MUA Alone | MUA With Dexamethasone and Celecoxib
Number analyzed (Participants) | 14 | 13
t-score
  6 weeks after MUA | 41.0 (5.3) | 42.5 (8.4)
  1 year after MUA: number analyzed (Participants) | 7 | 13
  1 year after MUA | 52.2 (6.2) | 45.2 (10.2)

14. Secondary Outcome: PROMIS-29 Outcome Form: Anxiety
Description: The PROMIS-29 outcome form measures physical and mental health outcomes for patients. Patients responded to 29 questions in seven categories: physical function, pain interference, depressive symptoms, anxiety, ability to participate in social activities, and sleep disturbance. Scores were scaled so that an average healthy person would score 50 points. A higher score represents more of what is being measured. For anxiety, lower scores indicate less anxiety.
  Patient questionnaire responses are scored using the PROMIS-29 scoring algorithm. Scores are scaled to a mean of 50 for a healthy reference population with a standard deviation of 10.
Time Frame: 6 weeks after MUA, and 1 year after MUA
Population: Patients who completed the PROMIS-29 survey and returned it.
Measure: Mean (Standard Deviation); unit: t-score
Arm/Group | MUA Alone | MUA With Dexamethasone and Celecoxib
Number analyzed (Participants) | 14 | 13
t-score
  6 weeks after MUA | 48.3 (9.4) | 48.9 (9.4)
  1 year after MUA: number analyzed (Participants) | 7 | 13
  1 year after MUA | 43.6 (6.1) | 45.5 (8.8)

15. Secondary Outcome: PROMIS-29 Outcome Form: Depression
Description: The PROMIS-29 outcome form measures physical and mental health outcomes for patients. Patients responded to 29 questions in seven categories: physical function, pain interference, depressive symptoms, anxiety, ability to participate in social activities, and sleep disturbance. Scores were scaled so that an average healthy person would score 50 points. A higher score represents more of what is being measured. For depression, lower scores indicate fewer depressive symptoms.
  Patient questionnaire responses are scored using the PROMIS-29 scoring algorithm. Scores are scaled to a mean of 50 for a healthy reference population with a standard deviation of 10.
Time Frame: 6 weeks after MUA, and 1 year after MUA
Population: Patients who completed the PROMIS-29 questionnaire and returned it.
Measure: Mean (Standard Deviation); unit: t-score
Arm/Group | MUA Alone | MUA With Dexamethasone and Celecoxib
Number analyzed (Participants) | 13 | 13
t-score
  6 weeks after MUA | 46.6 (9.4) | 48.7 (8.6)
  1 year after MUA: number analyzed (Participants) | 7 | 13
  1 year after MUA | 41.0 (0) | 46.8 (8.4)

16. Secondary Outcome: PROMIS-29 Outcome Form: Fatigue
Description: The PROMIS-29 outcome form measures physical and mental health outcomes for patients. Patients responded to 29 questions in seven categories: physical function, pain interference, depressive symptoms, anxiety, ability to participate in social activities, and sleep disturbance. Scores were scaled so that an average healthy person would score 50 points. A higher score represents more of what is being measured. For fatigue, lower scores indicate less fatigue.
  Patient questionnaire responses are scored using the PROMIS-29 scoring algorithm. Scores are scaled to a mean of 50 for a healthy reference population with a standard deviation of 10.
Time Frame: 6 weeks after MUA, and 1 year after MUA
Population: Patients who completed the PROMIS-29 survey and returned it.
Measure: Mean (Standard Deviation); unit: t-score
Arm/Group | MUA Alone | MUA With Dexamethasone and Celecoxib
Number analyzed (Participants) | 14 | 13
t-score
  6 weeks after MUA | 46.6 (8.7) | 48.2 (8.5)
  1 year after MUA: number analyzed (Participants) | 7 | 13
  1 year after MUA | 39.3 (7.2) | 41.5 (8.9)

17. Secondary Outcome: PROMIS-29 Outcome Form: Sleep Disturbance
Description: The PROMIS-29 outcome form measures physical and mental health outcomes for patients. Patients responded to 29 questions in seven categories: physical function, pain interference, depressive symptoms, anxiety, ability to participate in social activities, and sleep disturbance. Scores were scaled so that an average healthy person would score 50 points. A higher score represents more of what is being measured. For sleep disturbance, lower scores indicate less sleep disturbance.
  Patient questionnaire responses are scored using the PROMIS-29 scoring algorithm. Scores are scaled to a mean of 50 for a healthy reference population with a standard deviation of 10.
Time Frame: 6 weeks after MUA, and 1 year after MUA
Population: Patients who completed the PROMIS-29 survey and returned it.
Measure: Mean (Standard Deviation); unit: t-score
Arm/Group | MUA Alone | MUA With Dexamethasone and Celecoxib
Number analyzed (Participants) | 14 | 13
t-score
  6 weeks after MUA | 54.7 (9.7) | 57.4 (8.6)
  1 year after MUA: number analyzed (Participants) | 7 | 13
  1 year after MUA | 48.3 (9.4) | 48.0 (7.5)

18. Secondary Outcome: PROMIS-29 Outcome Form: Social Activities
Description: The PROMIS-29 outcome form measures physical and mental health outcomes for patients. Patients responded to 29 questions in seven categories: physical function, pain interference, depressive symptoms, anxiety, ability to participate in social activities, and sleep disturbance. Scores were scaled so that an average healthy person would score 50 points. A higher score represents more of what is being measured. For social activities, higher scores indicate a better ability to participate in social roles and activities.
  Patient questionnaire responses are scored using the PROMIS-29 scoring algorithm. Scores are scaled to a mean of 50 for a healthy reference population with a standard deviation of 10.
Time Frame: 6 weeks after MUA, and 1 year after MUA
Population: Patients who completed the PROMIS-29 survey and returned it.
Measure: Mean (Standard Deviation); unit: t-score
Arm/Group | MUA Alone | MUA With Dexamethasone and Celecoxib
Number analyzed (Participants) | 14 | 13
t-score
  6 weeks after MUA | 49.2 (8.2) | 51.5 (9.2)
  1 year after MUA: number analyzed (Participants) | 7 | 13
  1 year after MUA | 62.3 (4.7) | 56.1 (10.5)

19. Secondary Outcome: PROMIS-29 Outcome Form: Pain Interference
Description: The PROMIS-29 outcome form measures physical and mental health outcomes for patients. Patients responded to 29 questions in seven categories: physical function, pain interference, depressive symptoms, anxiety, ability to participate in social activities, and sleep disturbance. Scores were scaled so that an average healthy person would score 50 points. A higher score represents more of what is being measured. For pain interference, higher scores indicate more frequent interference in activities due to pain.
  Patient questionnaire responses are scored using the PROMIS-29 scoring algorithm. Scores are scaled to a mean of 50 for a healthy reference population with a standard deviation of 10.
Time Frame: 6 weeks after MUA, 1 year after MUA
Population: Patients who completed the PROMIS-29 survey and returned it.
Measure: Mean (Standard Deviation); unit: t-score
Arm/Group | MUA Alone | MUA With Dexamethasone and Celecoxib
Number analyzed (Participants) | 14 | 12
t-score
  6 weeks after MUA | 56.1 (9.7) | 58.2 (7.3)
  1 year after MUA: number analyzed (Participants) | 7 | 11
  1 year after MUA | 47.4 (7.2) | 56.7 (12.4)

ADVERSE EVENTS:
Time Frame: Adverse events were monitored throughout the study from the beginning of enrollment until both the 6-months post-manipulation under anesthesia and 1-year post-manipulation under anesthesia timepoints had been reached. Approximately 1 year.
Description: All sites conducted monitoring for adverse events.
Arm/Group | MUA Alone | MUA With Dexamethasone and Celecoxib
All-Cause Mortality (participants affected / at risk) | 0/59 | 0/72
Serious Adverse Events (participants affected / at risk) | 0/59 | 0/72
Other Adverse Events (participants affected / at risk) | 0/59 | 1/72
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MUA Alone (N=59) | MUA With Dexamethasone and Celecoxib (N=72)
Head Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Patient sustained a head injury resulting in a concussion and eye contusion while enrolled in the study. This was reported to the Data and Safety Monitoring Board and deemed unanticipated but not serious or related to the study procedure.

LIMITATIONS AND CAVEATS:
Participant dropout rates were higher than anticipated for in the initial enrollment calculations, and patient reported outcome surveys had low completion rates. As a result, the target of 90 power for results was not achieved for all study outcome metrics. Additional study is warranted regarding NSAID administration strategy for MUA patients in order to determine if NSAIDs can be useful in combatting the inflammatory cascade which is associated with arthrofibrosis and post TKA stiffness.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-06-08): https://cdn.clinicaltrials.gov/large-docs/35/NCT02739035/Prot_SAP_000.pdf
  • Informed Consent Form (2022-02-04): https://cdn.clinicaltrials.gov/large-docs/35/NCT02739035/ICF_001.pdf